CLINICAL TRIAL: NCT00075634
Title: A Phase I Study of Decitabine (NSC# 127716, IND# 50733) in Combination With Doxorubicin and Cyclophosphamide in the Treatment of Relapsed or Refractory Solid Tumors
Brief Title: Decitabine, Doxorubicin, and Cyclophosphamide in Treating Children With Relapsed or Refractory Solid Tumors or Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01807; NCI-2012-01807 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000347393; COG-ADVL0215; ADVL0215 (Other: COG Phase I Consortium); ADVL0215 (Other: CTEP); U01CA097452 (NIH)
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Recurrent Neuroblastoma; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Neuroblastoma | interventions — Decitabine; Doxorubicin; Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim

ARMS (1):
- Arm I (Experimental): PART A (solid tumor patients): Patients receive decitabine IV over 1 hour on days 0-6 and doxorubicin IV over 15 minutes and cyclophosphamide IV over 1 hour on day 7. Patients then receive filgrastim (G-CSF) subcutaneously (SC) beginning on day 8 and continuing until blood counts recover OR pegfilgrastim SC once on day 8 or 9*. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  PART B (neuroblastoma patients): Once the MTD is determined for part A, patients are treated as in part A at the MTD.
  Interventions: Drug: decitabine; Drug: doxorubicin hydrochloride; Drug: cyclophosphamide; Biological: filgrastim; Biological: pegfilgrastim; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Biological: pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; GCSF-SD01; Neulasta; SD-01 sustained duration G-CSF
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of decitabine when given together with doxorubicin and cyclophosphamide in treating children with relapsed or refractory solid tumors or neuroblastoma. Drugs used in chemotherapy, such as decitabine, doxorubicin, and cyclophosphamide, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of decitabine in combination with doxorubicin and cyclophosphamide in children with relapsed or refractory solid tumors or neuroblastoma.

II. Determine the toxic effects of this regimen in these patients. III. Determine whether decitabine induces tumor caspase-8 demethylation and expression in these patients.

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetics of low-dose decitabine in these patients. II. Determine the biological and clinical response in patients treated with this regimen.

III. Compare patterns of peripheral blood gene expression, using gene expression profiling, in patients before and after treatment with decitabine.

OUTLINE: This is a multicenter, dose-escalation study of decitabine.

PART A (solid tumor patients): Patients receive decitabine IV over 1 hour on days 0-6 and doxorubicin IV over 15 minutes and cyclophosphamide IV over 1 hour on day 7. Patients then receive filgrastim (G-CSF) subcutaneously (SC) beginning on day 8 and continuing until blood counts recover OR pegfilgrastim SC once on day 8 or 9*. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of decitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

NOTE: *For patients > 45 kg

PART B (neuroblastoma patients): Once the MTD is determined for part A, patients are treated as in part A at the MTD.

Patients are followed at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of either of the following:

  * Solid tumor (part A)

    * No lymphoma
  * Neuroblastoma (part B)

    * Original diagnosis may be based on elevated urine vanillylmandelic acid (VMA) and homovanillic acid (HVA) and bone marrow examination
    * Accessible disease by bone marrow aspirate or tumor biopsy

      * No laparotomy, thoracotomy, endoscopy, or craniotomy for biopsy
* No known curative therapy OR therapy proven to prolong survival with an acceptable quality of life available
* No known brain or spinal cord metastases
* No CNS tumors
* Performance status - Karnofsky 50-100% (patients 11 to 21 years of age)
* Performance status - Lansky 50-100% (patients ≤ 10 years of age)
* Parts A and B without bone marrow infiltration:

  * Absolute neutrophil count ≥ 1,000/mm^3
  * Platelet count ≥ 100,000/mm^3 (transfusion independent)
* Part B with bone marrow infiltration (i.e., tumor metastatic to bone marrow with granulocytopenia, anemia, and/or thrombocytopenia):

  * Absolute neutrophil count ≥ 750/mm^3
  * Platelet count ≥ 50,000/mm^3 (transfusion independent)
* Hemoglobin ≥ 8.0 g/dL (transfusion allowed)
* No sickle cell anemia
* Bilirubin ≤ 1.5 mg/dL
* ALT ≤ 5 times upper limit of normal
* No significant hepatic dysfunction that would compromise the tolerability of decitabine or interfere with study procedures or results
* Creatinine based on age as follows:

  * ≤ 0.8 mg/dL (5 years of age and under)
  * ≤ 1.0 mg/dL (6 to 10 years of age)
  * ≤ 1.2 mg/dL (11 to 15 years of age)
  * ≤ 1.5 mg/dL (16 to 21 years of age)
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min
* No significant renal dysfunction that would compromise the tolerability of decitabine or interfere with study procedures or results
* Shortening fraction ≥ 28% by echocardiogram
* Ejection fraction of ≥ 45% by MUGA
* No significant pulmonary dysfunction that would compromise the tolerability of decitabine or interfere with study procedures or results
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to agents used in this study
* No uncontrolled serious infection
* No significant end-organ dysfunction that would compromise the tolerability of decitabine or interfere with study procedures or results
* Recovered from prior immunotherapy
* At least 7 days since prior biologic therapy
* More than 1 week since prior growth factor therapy (2 weeks for pegfilgrastim)
* More than 2 weeks since prior epoetin alfa
* At least 6 months since prior autologous stem cell transplantation
* At least 6 months since prior allogeneic bone marrow transplantation

  * Patients must have full organ recovery and no evidence of graft-versus-host disease
* No concurrent immunomodulating agents
* No concurrent immunotherapy
* No concurrent biologic therapy
* No concurrent epoetin alfa
* Recovered from prior chemotherapy
* More than 2 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas)
* Prior total lifetime cumulative anthracycline dose ≤ 450 mg/m^2 of doxorubicin or equivalent
* No other concurrent chemotherapy
* No concurrent hydroxyurea
* Recovered from prior radiotherapy
* More than 2 weeks since prior local palliative small port radiotherapy
* More than 6 months since prior substantial bone marrow irradiation (e.g., cranio-spinal irradiation, total body irradiation, or hemi-pelvic irradiation)
* No concurrent radiotherapy
* No other concurrent anticancer therapy
* No other concurrent investigational agents
* Concurrent oral iron supplementation for patients with a known iron deficiency or a microcytic hypochromic anemia allowed

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2003-12; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
MTD of decitabine, based on incidence of DLT graded according to NCI CTCAE version 3.0 (Part A) | Up to 28 days
Caspase-8 expression in bone marrow or tumor biopsy samples (Part B) | Up to 28 days

SECONDARY OUTCOMES:
Objective response rate | Up to 56 days
  Confidence intervals will be reported in addition to the estimated response rates.
Percent of apoptotic cells as assessed by a TUNEL assay | Up to 1 year
  A sign test or other appropriate nonparametric test may be used to assess whether there was an increase in the percent of apoptotic cells after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rani George, Principal Investigator — COG Phase I Consortium
Locations (1):
- Children's Oncology Group, Arcadia, California, United States